CLINICAL TRIAL: NCT01465282
Title: A Randomized, Placebo-controlled, Phase IIb Study to Evaluate the Efficacy, Safety and Tolerability of 0.05%, 0.1% and 0.5% w/w Topical CT327 When Applied Twice Daily in Subjects With Psoriasis Vulgaris
Brief Title: Evaluation of the Efficacy, Safety and Toleration of CT327 Ointment in Patients With Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Creabilis SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT327-2003
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Psoriasis Vulgaris
Keywords: psoriasis vulgaris; topical ointment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.05% (w/w) CT327 ointment (Experimental): 0.05% (w/w) CT327 ointment applied BID for up to 8 weeks.
  Interventions: Drug: CT327 0.05%
- 0.1% (w/w) CT327 ointment (Experimental): 0.1% (w/w) CT327 ointment applied BID for up to 8 weeks.
  Interventions: Drug: CT327 0.1%
- 0.5% (w/w) CT327 ointment (Experimental): 0.5% (w/w) CT327 ointment applied BID for up to 8 weeks.
  Interventions: Drug: CT327 0.5%
- Placebo ointment (Placebo Comparator): Placebo ointment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CT327 0.05% — 0.05% CT327 (w/w) ointment
  Arms: 0.05% (w/w) CT327 ointment
Drug: CT327 0.1% — 0.1% CT327 (w/w) ointment
  Arms: 0.1% (w/w) CT327 ointment
Drug: CT327 0.5% — 0.5% CT327 (w/w) ointment
  Arms: 0.5% (w/w) CT327 ointment
Drug: Placebo — Placebo
  Arms: Placebo ointment

SUMMARY:
The purpose of this study is to evaluate the effectiveness of 3 dose strengths of CT327 ointment (0.05%, 0.1% and 0.05% w/w) compared to a placebo, when applied twice daily for up to 8 weeks, to the psoriatic plaques of patients with psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged at least 18 years.
* Stable psoriasis vulgaris

Exclusion Criteria:

* Subjects with guttate, erythrodermic, exfoliative or pustular psoriasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of CT327 ointment (0.05%, 0.1% and 0.5% w/w) compared with placebo ointment. | Week 8

SECONDARY OUTCOMES:
Local and systemic toleration | 8 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- United States (8):
  - Hotsprings, Arkansas
  - San Ramon, California
  - Bay City, Michigan
  - Fridley, Minnesota
  - South Euclid, Ohio
  - Portland, Oregon
  - San Antonio, Texas
  - Spanish Fork, Utah
- United Kingdom (5):
  - Birmingham
  - Cardiff
  - Glasgow
  - Manchester
  - Merseyside